CLINICAL TRIAL: NCT03935100
Title: A Prospective Randomised Placebo Controlled Trial on Prophylactic Endoscopic Clipping of Colonic Diverticula (PECoD)
Brief Title: Prophylactic Endoscopic Clipping of Diverticula (PECoD)
Acronym: PECoD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 253898
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Diverticular Disease
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinded to clipping, undergo same procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): All visible diverticula clipped during index colonoscopy
  Interventions: Procedure: Endoscopic clipping
- Control Group (Placebo Comparator): 5 clips fired at random into colon lumen. No diverticula closed.
  Interventions: Other: Placebo - colonoscopy without clipping

INTERVENTIONS:
Procedure: Endoscopic clipping — Endoscopic clips fired to close mucosa over diverticular defects.
  Arms: Treatment Group
Other: Placebo - colonoscopy without clipping — Colonoscopy performed, no clipping of diverticula
  Arms: Control Group

SUMMARY:
This study will evaluate the effect of endoscopic clipping of colonic diverticula in treatment of symptoms related to diverticular disease. Half of the participants will undergo colonoscopy without the clipping procedure and half will have colonoscopy with clipping of all visible diverticula.

DETAILED DESCRIPTION:
Colonic diverticular disease (DD) is characterised by the presence of sac-like protrusions (diverticula), which form through defects in the muscle layer of the colon wall. It is prevalent in western countries, affecting approximately 70% of individuals by the age of 80. The risk of acquiring diverticular disease increases uniformly with age, with approximately 40% of people aged over 60 years affected in western countries. Diverticular complications may be severe and include pain, inflammation, infection and bleeding. Although the majority of people with diverticular disease are asymptomatic, approximately 25% will experience an episode of acute diverticulitis (the principal inflammatory complication of diverticulosis); of these, 15% will develop other significant and often serious complications such as abscess, fistula or perforation.

King's College Hospital operates a tertiary referral service for patients with diverticular disease that integrates a gastroenterological and colorectal surgical approach to treatment. The investigators increasingly find that many patients have characteristic DD pain and IBS like symptoms with or without a clearly defined episode of diverticulitis. The link between symptomatic diverticular disease and Irritable Bowel Symptoms is reflected to some extent in the literature, however, it remains a matter of significant controversy. Nevertheless, these symptoms are often difficult to control and can be debilitating. Current treatment options for the IBS like symptoms in symptomatic uncomplicated DD are limited. In this age group, a low FODMAP diet, the mainstay treatment for IBS, is impractical and there are few if any controlled studies that address these issues. There is hence a need for alternative therapeutic options. Secondly, complications related to DD are associated with significant morbidity and mortality and comes at significant cost to the health service. At present there is no proven prophylactic intervention to prevent the complications.

The investigators have recently published the results of a feasibility study carried out at King's College Hospital, which assessed the effectiveness of elective endoscopic clipping of diverticula in patients with a history of significant diverticular bleeding. Here, all visible diverticula were closed endoscopically using 'Instinct' endoclips. A diverticula closure rate of 87.2% (129/148) was demonstrated at follow up colonoscopy. In this group, there were no post-procedural complications and no diverticula-associated symptoms reported up to the follow-up colonoscopy. Notably, incidental complete resolution of chronic left sided abdominal pain was noted in one of our subjects.

The investigators now propose the use of elective diverticular clipping in patients with symptomatic diverticulosis with a view to alter the natural history of the disease i.e. to prevent complications of the disease. At the same time the investigators wish to assess their symptomatic response. Patients with symptomatic diverticular disease will be eligible. The trial will be carried out at King's College Hospital endoscopy suite, a tertiary referral centre for endoscopic procedures. The study will include 84 patients. Each patient will be in the study for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed symptomatic diverticular disease (5 or more diverticula)
* Age range 18-90 years
* Retains capacity and medically fit for colonoscopy

Exclusion Criteria:

* Does not meet inclusion criteria
* Unable to give informed consent
* Patients with severe co-morbidities and substance misuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Rate of diverticula closure | 12 months
  Number of diverticula pre and post clipping

SECONDARY OUTCOMES:
Changes in abdominal symptoms | 12 months
  Changes in abdominal symptoms as assessed by the Irritable Bowel Syndrome Symptom Severity Score before and at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No